CLINICAL TRIAL: NCT06907147
Title: Global Pilot Study of rEnal and Hepatic coMbINed denervatIon in Subjects With Uncontrolled Hypertension With and Without High Cardiovascular Risk
Brief Title: SPYRAL GEMINI Pilot Study
Acronym: SPYRAL GEMINI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT23034
Record Dates: First submitted 2025-03-10; First posted 2025-04-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases; Chronic Kidney Diseases; Diabetes Mellitus
Keywords: Renal Insufficiency; Chronic Disease; Disease Attributes; Pathologic Processes; Kidney Diseases; Hypertension; Cardiovascular Diseases; Vascular Diseases; Denervation; Renal Denervation; Hepatic Denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus; Renal Insufficiency; Chronic Disease; Disease Attributes; Pathologic Processes; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Two parallel single-arm assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Gemini Pilot Off Med: Multi-Organ Denervation for Hypertension Off Anti-hypertensive Meds (Experimental)
  Interventions: Device: Multi-Organ Denervation Gemini System
- Gemini Pilot On Med: MDN for Hypertension and High Cardiovascular Risk On Anti-hypertensive Meds. (Experimental)
  Interventions: Device: Multi-Organ Denervation Gemini System

INTERVENTIONS:
Device: Multi-Organ Denervation Gemini System — After angiography according to standard procedures, subjects are treated with renal denervation followed by hepatic denervation.

SUMMARY:
The purpose of the SPYRAL GEMINI Pilot Study is to evaluate that multi-organ denervation with the Gemini System is safe and provide evidence of blood pressure reduction when studied in an uncontrolled hypertensive population with and without high cardiovascular risk.

DETAILED DESCRIPTION:
This study is exploratory in nature and will evaluate procedural and long-term safety of multi-organ denervation (MDN) and provide preliminary efficacy data in two parallel single arm cohorts:

* Gemini Pilot Off Med: MDN for Hypertension Off Anti-hypertensive Meds and,
* Gemini Pilot On Med: MDN for Hypertension and High Cardiovascular Risk On Anti-hypertensive Meds

There is no pre-specified primary endpoint; however, the data will be used for hypothesis generation to be evaluated and confirmed in subsequent clinical investigation(s).

ELIGIBILITY:
Inclusion Criteria:

All Subjects (both cohorts):

1. ≥18 and ≤80 years of age.
2. Diagnosed with HTN and has a baseline office SBP ≥150 mmHg and <180 mmHg and an office DBP ≥ 90 mmHg.
3. 24-hour average SBP ≥140 mmHg and <170 mmHg measured by ABPM at Baseline.

Exclusion Criteria:

1. Individual lacks appropriate renal artery OR common hepatic artery anatomy.
2. Prior renal or hepatic denervation.
3. Prior stroke or transient ischemic attack (TIA).
4. Documented Type 1 diabetes or use of insulin or sulfonylureas within 6 months.
5. Secondary cause of hypertension.
6. Documented condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement.
7. Estimated glomerular filtration rate (eGFR) of <40
8. Pregnant, nursing or planning to become pregnant during the study.
9. Primary pulmonary arterial hypertension.
10. History or evidence of active / suspected chronic liver or biliary disease.
11. Current or chronic pancreatitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-12-22 (Estimated); Study Completion 2029-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in office blood pressure | From baseline to 36 months post-procedure

OTHER OUTCOMES:
Change in 24-hour ambulatory blood pressure | From baseline to 3 and 6 months post-procedure
  Change in blood pressure from baseline as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) at 3-and 6-months post-procedure
Change in daytime blood pressure | From baseline to 3 and 6 months post-procedure
  Change in daytime blood pressure from baseline as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) at 3- and 6-months post-procedure
Change in nighttime blood pressure | From baseline to 3 and 6 months post-procedure
  Change in nighttime blood pressure from baseline as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) at 3- and 6-months post-procedure
Change in office blood pressure | From baseline to 1, 3, 6, 12, 24 and 36 months post-procedure
  Change in office blood pressure from baseline at 1-, 3-, 6-, 12-, 24- and 36-months post-procedure
Change in home blood pressure (HBP) | From baseline to 1, 3, 6, 12, 24 and 36 months post-procedure
  Change in home blood pressure (HBP) from baseline at 1-, 3-, 6-, 12-, 24- and 36-months post-procedure
Incidence of achieving target office systolic blood pressure (SBP<140 mmHg) | From baseline to 1, 3, 6, 12, 24 and 36 months post-procedure
  Incidence of achieving target office systolic blood pressure (SBP<140 mmHg) at 1-, 3-, 6-, 12-, 24- and 36-months post-procedure
All-cause mortality | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Significant embolic event resulting in end-organ damage | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Vascular complications | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Hospitalization for hypertensive crisis not related to non-adherence with medications or the protocol | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Major bleeding requiring transfusion | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Hepatic Arterial Damage requiring intervention (i.e., perforation, dissection, occlusion, aneurysm) | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Hepatic artery thrombosis | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
New Hepatic Stenosis >70%, confirmed by angiography | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Aminotransferase Elevation(s) >3x the upper limit of normal | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Myocardial Infarction | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Stroke | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Renal artery re-intervention | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
New renal artery stenosis >70% confirmed by angiography | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
End Stage Renal Disease or dialysis | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Increase in serum creatinine >50% from Baseline | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure
Any of the following requiring intervention or hospitalization: Pancreatitis, Biliary stricture, New onset biliary dyskinesia, Acute cholecystitis, Sphincter of Oddi dysfunction | From pre-procedure to immediately after the procedure, 1, 3, 6, 12, 24 and 36 months post-procedure

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - Stanford Hospital and Clinics, Stanford, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Providence Hospital, Southfield, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Renown Regional Medical Center, Reno, Nevada
  - Virtua Our Lady of Lourdes Hospital, Camden, New Jersey
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - UT Health East Texas, Tyler, Texas
- Royal Perth Hospital (Dobney Hypertension Centre), Perth, Australia
- Hippokration General Hospital, Athens, Greece
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.